CLINICAL TRIAL: NCT01403623
Title: A Randomized Trial to Evaluate the Use of Plastic Bags in Preventing and Treating Hypothermia in Neonates in Developing Countries
Brief Title: Evaluate the Use of Plastic Bags in Preventing and Treating Hypothermia in Neonates
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Alicia Leadford, MD, Fellow Instructor, Department of Pediatrics, Division of Neonatology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAB Neo 003
Record Dates: First submitted 2011-06-27; First posted 2011-07-27 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Hypothermia, Newborn
Keywords: Hypothermia; Newborn; Resuscitation; Plastic bag
MeSH Terms: conditions — Hypothermia | interventions — Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resuscitation with plastic bag (Active Comparator): Plastic bag will be used during and after resuscitation to assist with temperature regulation.
  Interventions: Procedure: Resuscitation and post resuscitation care with plastic bag
- Standard resuscitation- no plastic bag (Sham Comparator): Infant will be resuscitated per standard of care without being placed in a plastic bag for temperature regulation.
  Interventions: Procedure: Resuscitation- no plastic bag for temperature regulation

INTERVENTIONS:
Procedure: Resuscitation and post resuscitation care with plastic bag — Infant will be resuscitated and placed in a plastic bag up to his/her neck and around the back of his head (not covering the face) in the delivery room and taken to the nursery. The infant will remain in the plastic bag until first axillary temperature remains stable at 36.5-37.5 degrees Celsius. Expected length of time approximately one hour.
  Arms: Resuscitation with plastic bag
Procedure: Resuscitation- no plastic bag for temperature regulation — Infant will be resuscitated in the delivery room and taken to the nursery. The infant will be observed per unit standard until first axillary temperature remains stable at 36.5-37.5 degrees Celsius. Expected length of time approximately one hour.
  Arms: Standard resuscitation- no plastic bag

SUMMARY:
The overall hypothesis is that placing infants 1000-2500 grams in plastic bags when compared to routine care will reduce the risk of hypothermia (< 36.5 degrees C) without increasing hyperthermia (> 37.5 degrees C).

DETAILED DESCRIPTION:
Prevention

After consent, infants with estimated gestational age between 26-36.6 weeks or with expected birth weight 1000-2500 grams will be randomized to resuscitation per standard protocol or to resuscitation per standard protocol and plastic bag. The intervention group will be placed into a plastic bag covering the body and back and top of head (excluding face) prior to drying the body's surface. Resuscitation efforts continue per standard of care. The infant will remain in the bag through the admission process until his/her axillary temp is in the range of 36.5- 37.5 degrees Celsius. At this time, the bag will be discontinued and discarded. Standard temperature control will be continued per nursery standard. Skin-to-skin contact between mother and baby is not excluded; however, the infant will remain in the plastic bag. Infant's axillary temperature will be measured per nursery standard after discontinuation of plastic bag. The control group will receive standard of care thermoregulation. Secondary measures (i.e. blood pressures, glucose levels, weight gain, observation for respiratory distress syndrome, bronchopulmonary dysplasia, pneumothorax, sepsis, seizures, intraventricular hemorrhage, necrotizing enterocolitis, pulmonary hemorrhage, and death) will be recorded in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age 26-36.6 weeks or expected birth weight 1000-2500 grams.
* Delivery in the hospital.

Exclusion Criteria:

* Abdominal wall defect or myelomeningocele.
* Major congenital anomaly.
* Blistering skin disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Axillary temperature 36.5-37.5 degrees Celsius | 1-4 hours
  Temperature taken per axilla for 1 minute

SECONDARY OUTCOMES:
Blood pressure | Duration of hospitalization-expected average of 4 weeks
  Measure of extremity blood pressure per cuff taken during nursery stay.
Blood glucose | Duration of hospitalization-expected average of 4 weeks
  Measure of blood glucose per laboratory value taken per heelstick
Seizure | Duration of hospitalization-expected average of 4 weeks
  Seizure activity diagnosed by medical doctor or nurse. No electroencephalogram will be done.
Weight gain | Duration of hospitalization-expected average of 4 weeks
  Infant will be weighed daily and rates of weight gain will be measured.
Respiratory Distress Syndrome (RDS) | Duration of hospitalization-expected average of 4 weeks
  Documentation of increased work of breathing, retractions, and a need for oxygen, intubation, or surfactant.
Bronchopulmonary dysplasia (BPD) | 28 days after birth
  Oxygen requirement at 28 days of life
Pneumothorax | Duration of hospitalization-expected average of 4 weeks
  Either chest radiograph documentation or clinical deterioration consistent with air leak
Sepsis | Duration of hospitalization-expected average of 4 weeks
  Culture proven or culture negative clinically treated course consistent with sepsis.
Major brain injury | Duration of hospitalization-expected average of 4 weeks
  Intracranial hemorrhage Grade 3-4 or periventricular leukomalacia documented on cranial ultrasound
Necrotizing enterocolitis or intestinal perforation | Duration of hospitalization-expected average of 4 weeks
  Documentation of pneumatosis or intestinal perforation on x ray or treatment course for clinical necrotizing enterocolitis per Bell's stage greater than one.
Pulmonary hemorrhage | Duration of hospitalization-expected average of 4 weeks
  Blood seen in the endotracheal tube and treated by physician.
Death | Duration of hospitalization-expected average of 4 weeks
  Cardiorespiratory failure

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Study Director — University of Alabama at Birmingham; Alicia E Leadford, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

REFERENCES:
- [Derived] Leadford AE, Warren JB, Manasyan A, Chomba E, Salas AA, Schelonka R, Carlo WA. Plastic bags for prevention of hypothermia in preterm and low birth weight infants. Pediatrics. 2013 Jul;132(1):e128-34. doi: 10.1542/peds.2012-2030. Epub 2013 Jun 3. PMID 23733796